CLINICAL TRIAL: NCT03301662
Title: Transient Electrocardiogram Assessment in Stroke Evaluation
Acronym: TEASE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Region Gävleborg (Other)
Responsible Party: Sponsor
Other Study IDs: 2017321
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: atrial fibrillation; cryptogenic stroke; ECG screening; health-related quality of life; Short Form-36; stroke; thumb-ECG
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: chest and thumb- ECG — chest and thumb- ECG using the Coala Heart Monitor

SUMMARY:
In stroke survivors, atrial fibrillation is typically detected with short-term electrocardiogram (ECG) monitoring in the stroke unit. Prolonged continuous ECG monitoring is impractical and requires substantial resources while insertable cardiac monitors are invasive and costly. Chest and thumb-ECG could provide an alternative for atrial fibrillation detection post-stroke.

The primary objective of our study is to assess the incidence of newly diagnosed atrial fibrillation during 28 days of chest and thumb-ECG monitoring in patients with cryptogenic stroke. Secondary objectives are to assess Health-related Quality of Life using Short Form-36 and the feasibility of the Coala Heart Monitor in patients with stroke.

DETAILED DESCRIPTION:
Stroke survivors in Region Gävleborg, Sweden, will be eligible for the study from October 2017. Patients with a history of ischemic stroke without documented atrial fibrillation before or during ECG evaluation in the stroke unit will be evaluated by the chest and thumb-ECG system Coala Heart Monitor. The monitoring system is connected to a smart phone application which allows for remote monitoring and prompt advice on clinical management. Over a period of 28 days, patients will be monitored twice daily and may activate the ECG recording at symptoms. Upon completion, the system is returned by mail. This system offers a possibility to evaluate the presence of atrial fibrillation post-stroke, but the feasibility of this system in patients who recently suffered from a stroke is unknown. In addition Health-related Quality of Life using Short Form-36 in comparison to Swedish population norms will be assessed. The feasibility of the Coala Heart Monitor will be assessed by a self-developed questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged ≥18 years, with a validated diagnosis of ischemic cryptogenic stroke are eligible for the study.

Exclusion Criteria:

* For screening with chest and thumb-ECG, exclusion criteria are as follows: previously known atrial arrhythmia with an indication for anticoagulation, implantable defibrillator, pacemaker or insertable cardiac monitor, pregnancy, permanent indication for anticoagulation (including low-molecular weight heparin) due to atrial arrhythmia, mechanical heart valve, deep vein thrombosis, or pulmonary embolism. Patients with a life expectancy ≤6 months (e.g. severe heart failure New York Heart Association functional class IV or malignancy) are likewise excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinically confirmed diagnosis of ischemic stroke will be recruited from the catchment area of Region Gävleborg, Sweden. Eligible patients will be identified from daily checks of the medical records in the stroke unit. The recruitment is planned to start in October 2017.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-09 (Estimated); Primary Completion 2018-10-09 (Estimated); Study Completion 2019-10-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of atrial arrhythmia | 28 days (prospectively)
  Cumulative incidence of atrial arrhythmia at 28 days.

SECONDARY OUTCOMES:
Previous atrial arrhythmia | 10 years (retrospectively)
  The prevalence of previously known atrial arrhythmia before cryptogenic stroke and the number of these patients who had anticoagulant therapy.
Compliance with chest and thumb-ECG | 28 days (prospectively)
  Compliance with chest and thumb-ECG at week four (number of recorded scheduled ECG tracings).
Patient-reported experience with chest and thumb-ECG | 6 weeks (prospectively)
  Patient-reported experience with chest and thumb-ECG measured at week six
Health-related Quality of Life | 12 months prospectively
  Health-related Quality of Life (Short Form-36) at week 6 and at 12 months and the association with atrial fibrillation and compliance with chest and thumb-ECG.
Cumulative incidence of stroke | 3 years prospectively
  Cumulative incidence of stroke (and all-cause mortality) after three years in patients with atrial fibrillation versus without atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Hirsh M Koyi, MD PhD, Principal Investigator — Uppsala University/Region Gävleborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Result] Ruff CT, Giugliano RP, Braunwald E, Hoffman EB, Deenadayalu N, Ezekowitz MD, Camm AJ, Weitz JI, Lewis BS, Parkhomenko A, Yamashita T, Antman EM. Comparison of the efficacy and safety of new oral anticoagulants with warfarin in patients with atrial fibrillation: a meta-analysis of randomised trials. Lancet. 2014 Mar 15;383(9921):955-62. doi: 10.1016/S0140-6736(13)62343-0. Epub 2013 Dec 4. PMID 24315724
- [Result] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Result] Sjalander S, Sjalander A, Svensson PJ, Friberg L. Atrial fibrillation patients do not benefit from acetylsalicylic acid. Europace. 2014 May;16(5):631-8. doi: 10.1093/europace/eut333. Epub 2013 Oct 24. PMID 24158253
- [Result] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P, Agewall S, Camm J, Baron Esquivias G, Budts W, Carerj S, Casselman F, Coca A, De Caterina R, Deftereos S, Dobrev D, Ferro JM, Filippatos G, Fitzsimons D, Gorenek B, Guenoun M, Hohnloser SH, Kolh P, Lip GY, Manolis A, McMurray J, Ponikowski P, Rosenhek R, Ruschitzka F, Savelieva I, Sharma S, Suwalski P, Tamargo JL, Taylor CJ, Van Gelder IC, Voors AA, Windecker S, Zamorano JL, Zeppenfeld K. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Europace. 2016 Nov;18(11):1609-1678. doi: 10.1093/europace/euw295. Epub 2016 Aug 27. No abstract available. PMID 27567465
- [Result] Schnabel RB, Yin X, Gona P, Larson MG, Beiser AS, McManus DD, Newton-Cheh C, Lubitz SA, Magnani JW, Ellinor PT, Seshadri S, Wolf PA, Vasan RS, Benjamin EJ, Levy D. 50 year trends in atrial fibrillation prevalence, incidence, risk factors, and mortality in the Framingham Heart Study: a cohort study. Lancet. 2015 Jul 11;386(9989):154-62. doi: 10.1016/S0140-6736(14)61774-8. Epub 2015 May 7. PMID 25960110
- [Result] Andersson T, Magnuson A, Bryngelsson IL, Frobert O, Henriksson KM, Edvardsson N, Poci D. All-cause mortality in 272,186 patients hospitalized with incident atrial fibrillation 1995-2008: a Swedish nationwide long-term case-control study. Eur Heart J. 2013 Apr;34(14):1061-7. doi: 10.1093/eurheartj/ehs469. Epub 2013 Jan 14. PMID 23321349
- [Derived] Magnusson P, Lyren A, Mattsson G. Patient-reported feasibility of chest and thumb ECG after cryptogenic stroke in Sweden: an observational study. BMJ Open. 2020 Oct 28;10(10):e037360. doi: 10.1136/bmjopen-2020-037360. PMID 33115891
- [Derived] Magnusson P, Lyren A, Mattsson G. Diagnostic yield of chest and thumb ECG after cryptogenic stroke, Transient ECG Assessment in Stroke Evaluation (TEASE): an observational trial. BMJ Open. 2020 Sep 24;10(9):e037573. doi: 10.1136/bmjopen-2020-037573. PMID 32973062
- [Derived] Magnusson P, Koyi H, Mattsson G. A protocol for a prospective observational study using chest and thumb ECG: transient ECG assessment in stroke evaluation (TEASE) in Sweden. BMJ Open. 2018 Apr 3;8(4):e019933. doi: 10.1136/bmjopen-2017-019933. PMID 29615448